CLINICAL TRIAL: NCT03058107
Title: Tight Caloric Control in the Cachectic Oncologic Patient (TiCaCONCO or CoCooN) Can Stabilize Body Weight, Thereby Reducing Morbidity and Mortality: Validation of the Pilot Study - A Randomized Controlled Double-Blind Trial
Brief Title: Tight Caloric Control in the Cachectic Oncologic Patient (TiCaCONCO or CoCooN)
Acronym: TiCaCONCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Baxter Healthcare Corporation (Industry); Nutricia, Inc. (Industry)
Responsible Party: Principal Investigator, Elisabeth De Waele, MD, PhD, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUN 143201629790
Record Dates: First submitted 2017-01-10; First posted 2017-02-20 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Metabolism and Nutrition Disorder
Keywords: Nutrition Therapy
MeSH Terms: conditions — Nutrition Disorders | interventions — Nutrition Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Therapy (NT) group (Experimental): Nutrition Therapy is intensive dietary counseling based on practical measurements of energy expenditure, rather than calculating it using theoretic formulas or no method at all.
  Interventions: Dietary Supplement: Nutrition Therapy
- Control Therapy (CT) group (Active Comparator): Control Therapy is standard dietary counseling bij state-wide recognized onco-dietitians. Energy expenditure is never measured in this standard protocol.
  Interventions: Dietary Supplement: Control Therapy

INTERVENTIONS:
Dietary Supplement: Nutrition Therapy — At the time of diagnosis, patients will immediately be screened and started with Nutrition Therapy if assigned to group A. This regimen will stay in place for 6 weeks to 3 months, after which a switch will be made towards normal dietary counselling. Nutrition Therapy can be given orally, parenterally or via tube feeding (enteral nutrition), depending on the patient's status and aims at matching Caloric Intake with Resting Energy Expenditure. Moreover, a switch between these modalities is possible. Afterwards, standard dietary counselling will be given during the remainder of the study. Follow-up will last one year. If 6 months after the last enrolment the study shows a large difference with the control group, the study will be stopped for ethical reasons.
  Arms: Nutrition Therapy (NT) group
Dietary Supplement: Control Therapy — At the time of diagnosis, patients will immediately be screened and started with standard dietary counselling for 1 year if assigned to group B. Dietary intervention can be orally, parenterally or via tube feeding (enteral nutrition), depending on the patient's status. Moreover, a switch between these modalities is possible. Follow-up will last 1 year. If 6 months after the last enrolment the study shows a large difference with the control group, the study will be stopped for ethical reasons.
  Arms: Control Therapy (CT) group

SUMMARY:
Cancer is a worldwide spread disease with high prevalence and incidence, often of poor prognosis because it is typically diagnosed in an advanced stage. Another reason for this prognosis is the presence of malnutrition, on the one hand because of a diminished intake (due to anorexia), and on the other hand because of tumor-induced hypercatabolism. The result is a pathological state of the body called "cachexia", generally defined as a weight loss > 5% during the last 6 months before diagnosis. It had already been demonstrated that correct nutrition in such patients can limit morbidity, while promoting progression-free survival as well as well-being. The pilot study, previously performed by the investigators, was the first to suggest that Nutrition Therapy, based on the ESPEN guidelines and resting energy expenditure measured by indirect calorimetry, can promote overall survival. The aim of this project is to validate these preliminary results in a larger RCT (randomized controlled double-blind trial), to promote Nutrition Therapy as a novel modality in its own right in the treatment of cancer, rather than being merely supportive.

DETAILED DESCRIPTION:
In the investigators' pilot trial, 20 patients were randomized, 10 receiving regular counseling by regular oncodietitians, while the 10 others received nutrition therapy. In the latter group, an assessment of biophysical parameters was made (including the Bioelectrical Impedance Analysis or BIA for body composition), and the patients' Energy Expenditure was assessed using indirect calorimetry. Afterwards, the patients received nutrition therapy according to the ESPEN (European Society for Parenteral and Enteral Nutrition) guidelines. Supplementary interventions were made to match caloric intake to energy expenditure (the 'Tight Caloric' approach), using enteral and parenteral nutrition if indicated, by an intensive coaching and follow-up to continue this nutrition strategy (with dieticians even being "on call" after hours). While the study follow-up lasted 2 years, nutrition therapy was only performed during the first 3 months. The results were striking: apart from keeping their body weight in balance, the patients of the nutrition therapy group counted much less unexpected hospitalisation days and they clearly lived much longer .

This project targets the validation of these results on a large scale. For this study, patients with either colorectal adenocarcinoma, lung carcinoma, oesofageal carcinoma, gastric carcinoma, pancreatic carcinoma and head and neck cancer, due to the high prevalence of cachexia in these patients will be included. A weight loss can also occur during treatment, and does not need to be present at the start of the study. Patients will be randomized, and the study is intended to be be double-blinded, although this will be difficult to maintain in practice due to the nature of the treatment. The recruitment phase will last 2 years, keeping refusals and dropouts in mind. Follow-up will last 1 year after inclusion, although the actual nutrition therapy will again last only during therapy (3 months for chemotherapy, 6 weeks for radiotherapy): the period of active oncological treatment. An intermediate analysis is already made after 6 months of follow-up. In case survival is already statistically significant, the trial will be stopped for ethical reasons. In case of a positive result, the investigators want to implement nutrition therapy as a standard treatment in cachectic cancer patients in Belgium.

In case of a positive outcome (i.e. mere confirmation of our published results), the major advantage of nutrition therapy will be its relatively low cost while still affecting morbidity and mortality significantly. This can be practically achieved by redefining the dietician's task. The patient's own active participation in the decision making process is an important surplus in well-being and overall treatment. In combination with decreased morbidity and mortality the benefit of the patient can be found on every level.

Protocol Amendment dd 12/06/2017

Background:

Due to lack of patients with 5% weight loss in 6 months and, by consequence, very low inclusion rate, it was decided to amend the protocol. To achieve this, a special cooperation with the department of Radiotherapy was established. The service sees many patients who lose weight during radiotherapy, partly because of cancer-related cachexia, but mostly due to the mucositis caused by radiotherapy itself, losing > 10% of their initial body weight (at the start of their therapy). This is especially seen in cancers of head and neck, oesophagus and stomach. Radiotherapy is performed on working days and treatments typically last 5-7 weeks (depending on indication).

Amendment:

* Inclusion of patients with colorectal, lung and pancreatic cancer will be changed to: Inclusion of patients with lung, gastric, oesophageal, head and neck and pancreatic cancer
* 5% weight loss over the past 6 months will be changed to: patients with the aforementioned cancers where radiotherapy will be part of their treatment (or will be the entire treatment)
* Duration of intervention of 3 months will be changed to: duration of intervention for the entire period of radiotherapy
* After recalculation of statistical power, only 48 patients will be needed instead of 96. With correction for dropouts, this will become 60 patients instead of 120. This means 30 controls and 30 patients in the intervention group.
* The amendment will be added to the registration at clinicaltrials.gov.

The procedure and flowchart will remain unchanged. Analysis of the data will remain: in whole, per cancer and per sex (the latter two criteria requiring 60 patients in each group).

Protocol Amendment dd 19/09/2017

Background:

The study has seen much more inclusions and is running well thanks to the previous amendment. Due to a typo, the colorectal cancer group was unfortunately omitted. Also, the absolute difference of survival in the TiCaCo trial after one year was similar to that after the second year.

Amendment:

* Colorectal cancer patients are still to be included. Otherwise, nothing changes concerning inclusion criteria.
* The follow-up will be shortened from 2 years to one year.
* The amendment will be added to the registration at clinicaltrials.gov.

Protocol Amendment dd 05/02/2019

Background:

The study needs 48 inclusions that remain in the study until the end. However, the number of dropouts is too high, severely compromising the study's statistical power. Therefore, an inclusion surplus of 20 - 25% is required.

Amendment:

* The inclusion period will be expanded to 31/12/2019 or the inclusion of 60 patients (including dropouts), whichever is sooner.
* The amendment will be added to the registration at clinicaltrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Male and female
* Colorectal, lung, oesofageal, gastric, pancreatic or head and neck cancer before chemo- or radiotherapy is started (naive to treatment), but surgery may already have been performed OR relapse > 3 months after initial oncologic therapy
* Oncologic cachexia (undesired weight loss > 5% in less than 6 months), before or during treatment
* Written informed consent / ability to give informed consent

Exclusion Criteria:

* concomitant second malignancy
* uncertainty of diagnosis
* patient unfit for chemotherapy, radiotherapy or surgery
* palliative treatment or terminal patient (life expectancy < 3 months)
* patient already participating in another study
* Pregnancy / lactation
* Any other pathology present that causes the patient to be unfit for oncologic therapy (e.g. end-stage renal failure, severe COLD, severe heart failure)
* Unable to adhere to protocol instructions (e.g. language barrier)
* Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
overall survival (mortality) | 1 year
  Overall survival (OS) will be calculated for the whole group of NT vs Control (as calculated with statistical power), for men and women.

SECONDARY OUTCOMES:
hospitalisation | 1 year
  number of unexpected hospitalisation days
morbidity | 1 year
  SF36 questionnaire
weight stabilisation (kg) | 1 year
  The stabilisation of the patient's body weight at the end of the study will be measured on a scale (in kg).
body composition (%) | 1 year
  The BIA (bio-electric impedance analysis) will be performed at the beginning and the end of the study.
energy expenditure (Kcal) | 1 year
  Next to indirect calorimetry to asses resting energy expenditure, Sensewear technology will be used to assess the patient's total energy expenditure.
complete remission | 1 year
  To assess the possibility of cure, complete remission of disease will be assessed by computed tomography (routine examination).

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth De Waele, MD, PhD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] De Waele E, Mattens S, Honore PM, Spapen H, De Greve J, Pen JJ. Nutrition therapy in cachectic cancer patients. The Tight Caloric Control (TiCaCo) pilot trial. Appetite. 2015 Aug;91:298-301. doi: 10.1016/j.appet.2015.04.049. Epub 2015 Apr 22. PMID 25912786